CLINICAL TRIAL: NCT04433312
Title: Impact of Cancellation of Non-urgent Surgical Cases on Patients During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa shalaby, MD, MSc, PhD, Dr, Mansoura University
Other Study IDs: SURG RES COL 2
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Satisfaction, Patient; Quality of Life
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The questionnaire is developed based on a literature review and clinical experience. Initial testing of the questionnaire will be performed with 20 patients to assess the reliability and inter-rater variations. After initial testing, the final questionnaire will be formulated. The first sector of the questionnaire includes patient demographics and baseline characteristics; the second sector is regarding patient clinical condition, diagnosis, and scheduled surgery. The following sector examines the process of delivering the cancellation to the patient and requirements for re-scheduling. Patients will be classified into satisfied or dissatisfied according to the responses in this sector. The following sector addresses the course of care after cancellation and whether the patient conducted the surgery elsewhere or not. The last sector explores the impact of cancellation on patient health, career, and financial aspects.

SUMMARY:
A questionnaire is developed based on the literature and clinical experience. Initial testing will be performed on 20 patients. The first and second sectors include patient demographics and patient clinical diagnosis/scheduled surgery, respectively. The following sectors examine the process of delivering the cancellation/re-scheduling; care after cancellation and whether the procedure conducted elsewhere or not; and the impact of cancellation on patient health, career, and financial aspects.

DETAILED DESCRIPTION:
This study is a cross-sectional survey of patients who were scheduled for elective surgical procedures and their surgeries were cancelled or postponed during the first wave of COVID-19 pandemic. The survey consists of a semi-structured questionnaire that is provided in the English language. A subsequent translation in patients' own Language will be provided based on geographical distribution. The survey will be conducted online, via email, or via telephone call based on the available and best method of participation according to involved hospital. Participants will be aware of the nature of the study and informed that their participation will be voluntary. Collected data will be confidential and anonymous.

The questionnaire is developed based on a literature review and clinical experience. Initial testing of the questionnaire will be performed with 20 patients to assess the reliability and inter-rater variations. Ambiguous questions and questions with a high rate of "I do not know" the answer will be excluded. To ensure high compliance, the questionnaire included the least possible number of questions. The questionnaire consists of closed questions except for two open questions that explore patients' suggestions to decrease the insult of cancellation on his life.

After initial testing, the final questionnaire will be formulated. The first sector of the questionnaire includes patient demographics and baseline characteristics; the second sector is regarding patient clinical condition, diagnosis, and scheduled surgery. The following sector examines the process of delivering the cancellation to the patient and requirements for re-scheduling. Patients will be classified into satisfied or dissatisfied according to the responses in this sector. The following sector addresses the course of care after cancellation and whether the patient conducted the surgery elsewhere or not. The last sector explores the impact of cancellation on patient health, career, and financial aspects. The impact of cancellation on patients' life will be classified into negative/positive/neutral based on the answers to this sector.

Statistical analyses will be performed using SPSS v. 20. Data distribution will be tested for normality using the Kolmogorov-Smirnov test and the Shapiro-Wilk test. Categorical variables will be expressed as group percentages and will be compared for independent samples using the Chi-square test. Continuous data of the survey will be presented as medians with ranges or means and standard deviations. A comparison of continuous data will be compared for independent samples using the T-test or Mann-Whitney test according to the data distribution. Spearman correlation coefficient will be used for further assessment of the strength of the association between variables. The statistical significance level will be set at <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Patients their elective surgeries were cancelled or postponed due to COVID-19 pandemic

Exclusion Criteria:

* Patients underwent surgery during COVID-19
* Emergency Surgeries

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Both sex
  * Patients their elective surgeries were cancelled or postponed due to COVID-19 pandemic
  * World wide
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life of the patients | During the COVID-19 pandemic 6 months (March-October 2020)
  A questionnaire based on the literature review to access the quality of the life of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Shalaby, MD, MSc, PhD, Principal Investigator — Mansoura University; Hosam Hamed, MD, MSc, PhD, Study Chair — Mansoura University; Ahmed M Elsheikh, MD,MBA,CMQOE, Study Director — Mansoura University
Locations (1):
- Mansoura Faculty of Medicine, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No